CLINICAL TRIAL: NCT06372067
Title: Intramedullary Screw Versus Kirschner Wire Fixation of Extraarticular Proximal and Middle Phalanx Fractures: Pilot Study for a Randomized Controlled Trial
Brief Title: IM Screw vs. K-wire Fixation of Proximal/Middle Phalanx Fractures
Acronym: HANDFIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Helene Retrouvey, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17378
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Hand; Fracture, Phalanx
MeSH Terms: conditions — Fractures, Bone | interventions — Bone Wires

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, pilot randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: By nature of the interventions in this study, blinding will not be possible for the surgeon or the patient post-operatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramedullary screw (Experimental): Intramedullary (IM) screw fixation is a minimally invasive technique that provides rigid fixation of fractures, acting as an internal splint and load-sharing device. IM screw fixation may allow for early mobilization without the operative site morbidity of open reduction and its associated complications.
  Interventions: Device: Intramedullary screw
- Kirschner wire (Active Comparator): Kirschner wire (K-wire) fixation is a minimally invasive technique that provides non-rigid fixation of fractures. K-wires allow for fracture fixation with minimal soft tissue injury and preserved blood supply. However, patients require prolonged postoperative immobilization and are at risk of malunion and pin tract infection.
  Interventions: Device: Kirschner wire

INTERVENTIONS:
Device: Intramedullary screw — Intramedullary (IM) screw fixation is a minimally invasive technique that provides rigid fixation of fractures, acting as an internal splint and load-sharing device. IM screw fixation may allow for early mobilization without the operative site morbidity of open reduction and its associated complications.
  Arms: Intramedullary screw
Device: Kirschner wire — Kirschner wire (K-wire) fixation is a minimally invasive technique that provides non-rigid fixation of fractures. K-wires allow for fracture fixation with minimal soft tissue injury and preserved blood supply. However, patients require prolonged postoperative immobilization and are at risk of malunion and pin tract infection.
  Arms: Kirschner wire

SUMMARY:
When people break their fingers, sometimes surgery is needed to align the bones to heal them properly. There are different ways to fix broken bones in hands, such as plates, pins, or screws. Each method has pros and cons; fixing a broken bone with plates is usually a larger surgery with more cutting but holds the bones very securely. Pins require little to no cutting but the patient needs to immobilize their hand for a few weeks afterwards. Screws are a newer method of fixing broken fingers that requires little cutting and also holds the bones securely. The goal of this study is to compare the effectiveness of using pins versus screws in surgery for broken fingers. The investigators are studying whether using screws leads to better hand function, patient satisfaction, and quicker return to work.

DETAILED DESCRIPTION:
Hand fractures are one of the most common skeletal injuries and affect a wide range of the population. Commonly affected groups include children and young adults with sports-related injuries, manual labourers with work-related injuries, and the elderly. Although the majority of phalanx fractures may be managed conservatively with good outcomes, operative fixation is indicated for significantly displaced or unstable fracture patterns, and those causing malrotation and scissoring.

There are a variety of options for operative fixation of proximal and middle phalanx fractures, which include closed versus open reduction (CR vs OR) with percutaneous pinning (PP) or internal fixation (IF) techniques. Kirschner wires (K-wire) and plates/screws are the most common CRPP and ORIF techniques. K-wires allow for fracture fixation with minimal soft tissue injury and preserved blood supply. However, patients require prolonged postoperative immobilization and are at risk of malunion and pin tract infection. Conversely, ORIF with plates/screws provide rigid fixation allowing for early mobilization, but require opening of fracture site and often periosteal stripping. Complications with ORIF include adhesions and stiffness.

There is emerging evidence for the effectiveness of intramedullary (IM) screw fixation as an alternative technique for IF. IM screw fixation is a minimally invasive technique that provides rigid fixation of fractures, acting as an internal splint and load-sharing device. Its biomechanical properties have been well-described in the lower extremity orthopedic literature. IM screw fixation may allow for early mobilization without the operative site morbidity of open reduction and its associated complications. Small observational cohort studies have shown favourable outcomes in return to activity, range of motion, time to radiological healing, and grip strength. However, the investigators' literature search revealed a paucity of high quality studies comparing the effectiveness of IM screws with K-wires or other methods of fixation.

The primary objective of this pilot study is to assess the feasibility of a randomized controlled trial comparing two CR techniques, i.e. IM screw fixation to K-wire fixation, in adult patients with extraarticular proximal or middle phalanx fracture at the investigators' tertiary academic hospital. The secondary objective will be to describe early clinical outcomes which can be used for future trial sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients ≥18 years old
2. scheduled for operative management of extraarticular proximal or middle closed phalanx fracture(s) at the investigators' tertiary hospital
3. feasible to perform closed reduction
4. able to provide informed consent and complete health-related quality of life (HRQoL) questionnaires in English

Exclusion Criteria:

1. other fractures that cannot be managed with IM screws or K-wires
2. other intraarticular fractures
3. significant concomitant hand trauma
4. cannot commit to 3 months of follow up at the investigators' institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patient Eligibility - Study Feasibility | 1 year
  The percentage of patients that are eligible for the study among those that are screened will be recorded. This criteria will be determined to be feasible if at least 70% of screened patients are deemed to be eligible.
Recruitment rate - Study Feasibility | 1 year
  The percentage of patients that are enrolled in the study among those determined to be eligible will be recorded. To be considered fully enrolled patients must sign the informed consent form, complete baseline demographic questionnaires, and be randomized to a study arm. This criteria will be determined to be feasible if at least 70% of eligible patients are recruited.
Crossover rate - Study Feasibility | 1 year
  The percentage of patients that crossover to the other arm of the study among those who are eligible and recruited for the study. This criteria will be determined to be feasible if no more than 5% of patients cross over.
Compliance with intervention rate - Study Feasibility | 1 year
  The percentage of patients that comply with the intervention (appropriate post-operative care, follow-up appointments) among those who are eligible and recruited for the study. This criteria will be determined to be feasible if at least 90% of patients are compliant.
Patient retention rate - Study Feasibility | 1 year
  The percentage of patients that complete patient-reported questionnaire (Disabilities of the Arm, Shoulder, and Hand) at the 3-month mark, which will be the primary outcome of the main trial. Scores range from 0-100 points, where higher scores indicate greater disability. This criteria will be determined to be feasible if at least 80% of patients are compliant.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder, and Hand | baseline, 4 weeks, 12 weeks
  The Disability of the Arm, Shoulder, and Hand is a region-specific PROM that has been shown to be valid, reliable, and responsive to change in measuring patient-important domains pertaining to the upper extremity. Scores range from 0-100 points, where higher scores indicate greater disability. In trauma populations, the Disability of the Arm, Shoulder, and Hand has been shown to have excellent internal consistency (0.98) and test-retest probability (intraclass correlation coefficient [ICC] = 0.98). The Disability of the Arm, Shoulder, and Hand has also been reported to have good criterion validity, construct validity and responsiveness in hand trauma patients.
Range of motion | 4 weeks, 8 weeks, 12 weeks
  Range of motion of the affected finger, compared to the contralateral finger. As measured and reported by hand therapist appointments which are part of routine care at the investigators' institution.
Grip strength | 8 weeks, 12 weeks
  Grip strength of the affected hand, compared to the contralateral hand. As measured and reported by hand therapist appointments which are part of routine care at the investigators' institution.
Return to work | through study completion, an average of 3 months
  Time of patient-reported return to work or surgeon clearance for return to work.
Complications/adverse events | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Post-operative complications/adverse events include but are not limited to stiffness, delayed union, non-union, malunion, infection, hardware removal, reoperation.
Postoperative pain (visual analogue scale) | 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Pain will be measured postoperative on the visual analogue scale, which ranges from 0-10. Higher scores indicate greater pain.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individualized participant data will not be shared.

REFERENCES:
- [Background] Meals C, Meals R. Hand fractures: a review of current treatment strategies. J Hand Surg Am. 2013 May;38(5):1021-31; quiz 1031. doi: 10.1016/j.jhsa.2013.02.017. PMID 23618458
- [Background] Kremer L, Frank J, Lustenberger T, Marzi I, Sander AL. Epidemiology and treatment of phalangeal fractures: conservative treatment is the predominant therapeutic concept. Eur J Trauma Emerg Surg. 2022 Feb;48(1):567-571. doi: 10.1007/s00068-020-01397-y. Epub 2020 May 25. PMID 32451567
- [Background] Gaio NM, Kruse LM. Closed Reduction Percutaneous Pinning Versus Open Reduction With Plate and Screw Fixation in Management of Unstable Proximal Phalangeal Fractures: A Systematic Review and Meta-analysis. Hand (N Y). 2025 Jan;20(1):136-142. doi: 10.1177/15589447231189762. Epub 2023 Aug 20. PMID 37599408
- [Background] Chao J, Patel A, Shah A. Intramedullary Screw Fixation Comprehensive Technique Guide for Metacarpal and Phalanx Fractures: Pearls and Pitfalls. Plast Reconstr Surg Glob Open. 2021 Oct 26;9(10):e3895. doi: 10.1097/GOX.0000000000003895. eCollection 2021 Oct. PMID 34712548
- [Background] Bong MR, Kummer FJ, Koval KJ, Egol KA. Intramedullary nailing of the lower extremity: biomechanics and biology. J Am Acad Orthop Surg. 2007 Feb;15(2):97-106. doi: 10.5435/00124635-200702000-00004. PMID 17277256
- [Background] del Pinal F, Moraleda E, Ruas JS, de Piero GH, Cerezal L. Minimally invasive fixation of fractures of the phalanges and metacarpals with intramedullary cannulated headless compression screws. J Hand Surg Am. 2015 Apr;40(4):692-700. doi: 10.1016/j.jhsa.2014.11.023. Epub 2015 Feb 7. PMID 25661294
- [Background] Patankar H, Meman FW. Multiple intramedullary nailing of proximal phalangeal fractures of hand. Indian J Orthop. 2008 Jul;42(3):342-6. doi: 10.4103/0019-5413.39573. PMID 19753163
- [Background] Verver D, Timmermans L, Klaassen RA, van der Vlies CH, Vos DI, Schep NWL. Treatment of extra-articular proximal and middle phalangeal fractures of the hand: a systematic review. Strategies Trauma Limb Reconstr. 2017 Aug;12(2):63-76. doi: 10.1007/s11751-017-0279-5. Epub 2017 Mar 4. PMID 28260179
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Deshmukh SR, Mousoulis C, Marson BA, Grindlay D, Karantana A; Core Outcome Set for Hand Fractures and Joint Injuries in Adults Group*. Developing a core outcome set for hand fractures and joint injuries in adults: a systematic review. J Hand Surg Eur Vol. 2021 Jun;46(5):488-495. doi: 10.1177/1753193420983719. Epub 2021 Jan 24. PMID 33487059
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Background] Ziebart C, Bobos P, Furtado R, Dabbagh A, MacDermid J. Patient-reported outcome measures used for hand and wrist disorders: An overview of systematic reviews. J Hand Ther. 2023 Jul-Sep;36(3):719-729. doi: 10.1016/j.jht.2022.10.007. Epub 2023 Mar 11. PMID 36914499
- [Background] Esteban-Feliu I, Gallardo-Calero I, Barrera-Ochoa S, Lluch-Bergada A, Alabau-Rodriguez S, Mir-Bullo X. Analysis of 3 Different Operative Techniques for Extra-articular Fractures of the Phalanges and Metacarpals. Hand (N Y). 2021 Sep;16(5):595-603. doi: 10.1177/1558944719873144. Epub 2019 Sep 13. PMID 31517524